CLINICAL TRIAL: NCT04049552
Title: Effect of Topical Rapamycin Ointment on Keloid Regression: A Pilot Study in Human Subjects (RAPA-Keloid)
Brief Title: RAPA-Keloid Study of Keloid Regression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20190291H
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Sirolimus; Ointments

STUDY DESIGN:
Intervention Model Description: Study participants will serve as their own control, using intervention on one keloid and placebo on the other
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RAPA intervention (Experimental): Rapamycin ointment will be applied to one keloid on the subject
  Interventions: Drug: Rapamycin 8% Ointment
- Placebo (Placebo Comparator): Placebo will be applied as a control on one keloid on the subject
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapamycin 8% Ointment — A compounded ointment containing 8% rapamycin
  Other Names: Rapamycin ointment
  Arms: RAPA intervention
Drug: Placebo — Petrolatum ointment placebo
  Other Names: Petrolatum ointment
  Arms: Placebo

SUMMARY:
1. To test whether topical rapamycin regresses established keloids in humans by measuring surface area and height changes in the scar over time (6 months)
2. To test safety of product and feasibility of conduct for future clinical trial

DETAILED DESCRIPTION:
This pilot trial will use daily 0.5-1.0 ml applications of 8% RAPA (Rapamycin) in a petrolatum vehicle to treat established keloid lesions in 5 persons with at least 2 chronic keloids in similar body regions (greater than 1-year duration). Treatment will be applied once daily for 6 months. One keloid will receive 8% RAPA ointment and the other keloid will receive petrolatum-only ointment as a control. Surface areas and height of keloids will be monitored pre- and post-treatment to evaluate responses.

Keloid surface area and height changes will be measured pre-treatment and thereafter on a monthly basis using standardized digital photography with a tripod-mounted 8MP Canon S5is camera and calipers to measure keloid height (37).

Surface areas of all photographed lesions will be measured with Image J (http://rsbweb.nih.gov/ij/index.html), a public image-processing program that was used to analyze preliminary data and this study will use the same approach.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have at least 2 keloid scars (for at least 1 year) in similar body locations that are easy to reach to apply ointment to
* Subject will be in good health with all chronic diseases (such as hypertension, coronary artery disease, etc.) clinically stable
* Cognitive functioning sufficient to provide informed consent
* Physically able to apply ointment to keloids daily
* Able to attend monthly clinic visits for 6 months

Exclusion Criteria:

* Diagnosis of diabetes
* Subjects taking the following medications: systemic steroid or immunosuppressant therapy within the past 6 months
* Local area steroidal treatment within the past 3 months
* History of allergy to rapamycin of petrolatum-based products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2021-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean L Kellogg Jr, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Audie L Murphy Memorial Veterans Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each subject enrolled was used as both active intervention and placebo, using 2 keloids on the same subject, color coded to have either rapamycin ointment or placebo ointment applied.
Units Other Than Participants: Keloids
Groups:
- Overall Study Participants: Rapamycin ointment will be applied to one keloid on the subject, and placebo will be applied to the second keloid on that subject. Keloids will be color coded to match either rapamycin ointment or placebo.
  Rapamycin 8% Ointment: A compounded ointment containing 8% rapamycin Placebo: Petrolatum ointment
Period: Overall Study
Arm/Group | Overall Study Participants
Started | 4; 8 Keloids
Completed | 3; 6 Keloids
Not Completed | 1; 2 Keloids
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Participants, each with 2 keloids, served as their own control, with one keloid color coded for active drug and the other for placebo
Units Other Than Participants: Keloids
Groups:
- Overall Study Participants: Rapamycin ointment will be applied to one keloid on the subject and placebo will be applied to a second keloid.
  Keloids will be color coded to match ointment applied
  Rapamycin 8% Ointment: A compounded ointment containing 8% rapamycin Placebo: Petrolatum ointment
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 3
Number analyzed (Keloids) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Keloid Surface Area
Description: Measurement of surface area of keloid
Time Frame: Baseline to 6 months
Measure: Mean (Full Range); unit: cm2
Units Other Than Participants: keloids
Arm/Group | RAPA Intervention | Placebo
Number analyzed (Participants) | 3 | 3
Number analyzed (keloids) | 3 | 3
cm2 | 0.455 [0.131 to 0.735] | -0.039 [-0.09 to -0.0075]

2. Secondary Outcome: Change in Keloid Height
Description: Measurement of height of keloid
Time Frame: Baseline to 6 months
Measure: Mean (Full Range); unit: millimeters
Units Other Than Participants: keloids
Arm/Group | RAPA Intervention | Placebo
Number analyzed (Participants) | 3 | 3
Number analyzed (keloids) | 3 | 3
millimeters
  Baseline | 1.5 [1.08 to 2.04] | 1.55 [1.29 to 1.93]
  6 months | 1.056 [0.4 to 1.54] | 0.93 [0.33 to 1.30]

ADVERSE EVENTS:
Time Frame: Baseline to 6 months.
Description: Any study related adverse event
Arm/Group | RAPA Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04049552/Prot_SAP_000.pdf